CLINICAL TRIAL: NCT00000549
Title: Estrogen Replacement and Atherosclerosis (ERA) in Older Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 93; U01HL049488 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases; Myocardial Ischemia; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Estrogen Replacement Therapy; Hormone Replacement Therapy; Estrogens; Progestins

INTERVENTIONS:
Drug: estrogen replacement therapy
Drug: hormone replacement therapy
Drug: estrogens
Drug: progestins

SUMMARY:
To determine if estrogen replacement therapy, with or without low dose progesterone, slows progression or induces regression of coronary atherosclerosis in postmenopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease is the number one cause of death in postmenopausal women. Postmenopausal estrogen replacement is associated with a lower incidence of cardiovascular disease in women, especially in those with established coronary artery disease. The strength of the apparent effect of estrogen in epidemiologic studies suggests that estrogen plays a fundamental role in the maintenance of vascular health. Animal data suggest that the current practice of adding the low dose progesterone to prevent endometrial hyperplasia may inhibit the beneficial effects of estrogen on coronary arteries. Before committing millions of postmenopausal women to long-term estrogen use for prevention of coronary artery disease, it is mandatory to demonstrate that it does indeed protect against coronary atherosclerosis, to determine the impact of co-treatment with progestin, and to understand the mechanisms through which estrogen may exert it's cardioprotective effects.

The Office of Research on Women's Health provided $500,000 in Fiscal Year 1995 for recruitment of subjects.

DESIGN NARRATIVE:

Randomized, placebo-controlled, blinded. The minimum diameter of coronary stenotic lesions was measured by angiography before and after three years in a group receiving unopposed estrogen replacement therapy, a group receiving estrogen replacement plus continuous low dose progestin, and a group receiving placebo. The incidence of clinical events was documented in all three groups. Secondary objectives of the trial included examining the effect of chronic and acute estrogen administration on endothelium-dependent coronary vasodilator capacity, plasma lipids and lipoproteins, antioxidant activity, blood pressure, glucose metabolism, and plasma hemostatic factors, as well as on behaviors, physical attributes, and psychosocial parameters. There were four pre-randomization variables in order to pre-stratify. These included current smoking status, insulin dependent diabetes, current lipid-lowering therapy, and the hospital where angiograms were performed.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women with established coronary atherosclerosis.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-08; Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Herrington — Bowman Gray School of Medicine

REFERENCES:
- [Background] Herrington DM, Reboussin DM, Klein KP, Sharp PC, Shumaker SA, Snyder TE, Geisinger KR. The estrogen replacement and atherosclerosis (ERA) study: study design and baseline characteristics of the cohort. Control Clin Trials. 2000 Jun;21(3):257-85. doi: 10.1016/s0197-2456(00)00054-4. PMID 10822123
- [Background] Folmar S, Oates-Williams F, Sharp P, Reboussin D, Smith J, Cheshire K, Macer J, Potvin Klein K, Herrington D. Recruitment of participants for the Estrogen Replacement and Atherosclerosis (ERA) trial. a comparison of costs, yields, and participant characteristics from community- and hospital-based recruitment strategies. Control Clin Trials. 2001 Feb;22(1):13-25. doi: 10.1016/s0197-2456(00)00117-3. PMID 11165419
- [Background] Herrington DM, Reboussin DM, Brosnihan KB, Sharp PC, Shumaker SA, Snyder TE, Furberg CD, Kowalchuk GJ, Stuckey TD, Rogers WJ, Givens DH, Waters D. Effects of estrogen replacement on the progression of coronary-artery atherosclerosis. N Engl J Med. 2000 Aug 24;343(8):522-9. doi: 10.1056/NEJM200008243430801. PMID 10954759
- [Background] Erkkila AT, Lichtenstein AH, Mozaffarian D, Herrington DM. Fish intake is associated with a reduced progression of coronary artery atherosclerosis in postmenopausal women with coronary artery disease. Am J Clin Nutr. 2004 Sep;80(3):626-32. doi: 10.1093/ajcn/80.3.626. PMID 15321802
- [Background] Herrington DM, Howard TD, Hawkins GA, Reboussin DM, Xu J, Zheng SL, Brosnihan KB, Meyers DA, Bleecker ER. Estrogen-receptor polymorphisms and effects of estrogen replacement on high-density lipoprotein cholesterol in women with coronary disease. N Engl J Med. 2002 Mar 28;346(13):967-74. doi: 10.1056/NEJMoa012952. PMID 11919305
- [Background] Lakoski SG, Brosnihan B, Herrington DM. Hormone therapy, C-reactive protein, and progression of atherosclerosis: data from the Estrogen Replacement on Progression of Coronary Artery Atherosclerosis (ERA) trial. Am Heart J. 2005 Nov;150(5):907-11. doi: 10.1016/j.ahj.2004.11.025. PMID 16290959